CLINICAL TRIAL: NCT06205043
Title: Enhancing Deep Brain Stimulation Programming for Parkinson's Disease: A Semi- Automatic Algorithm-Guided Approach Using StimSearch- A Double Blind Randomized Study
Brief Title: Algorithm Guided DBS Programming in Parkinson's Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaslok Hospital and Research Centre (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Paresh doshi, Director of Neurosurgery and Stereotactic and Functional Neurosurgical program, Jaslok Hospital and Research Centre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Stimulation Search
Record Dates: First submitted 2023-11-28; First posted 2024-01-12 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: Deep brain stimulation; Programming; Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either an algorithm based program vs standard of care program. After a period each group will cross over to the other side. UPDRS assessments will be done at each time.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of care (SoC) based programming in Parkinson's disease patients (Active Comparator): Patients will be programmed in a routine (Standard of Care) program. Based on the randomization the patient may receive this at the beginning or after the Stim search program (crossover)
  Interventions: Device: Clinician based programming
- StimSearchTM software based programing in Parkinson's disease patients (Experimental): Patients will be programmed using StimSearch algorithm. Based on the randomization the patient may receive this at the beginning or after the Standard of Care program (crossover)
  Interventions: Device: StimSearch programming algorithm software

INTERVENTIONS:
Device: StimSearch programming algorithm software — This is an algorithm based method to program deep brain stimulation in patients of Parkinson's disease
  Arms: StimSearchTM software based programing in Parkinson's disease patients
Device: Clinician based programming — This is Standard of Care programming performed for patients undergoing deep brain stimulation for Parkinson's disease
  Arms: Standard of care (SoC) based programming in Parkinson's disease patients

SUMMARY:
Patients undergoing Deep Brain Stimulation for Parkinson's disease will be subjected to standard of care programming and compared with the algorithm based programming (StimSearch). Various parameters including the effectivity and efficiency of algorithm programming will be compared against the standard of care programming.

DETAILED DESCRIPTION:
Patients of Parkinson's disease undergoing bilateral subthalamic nucleus stimulation (STN), we have already been adequately programmed and have achieved good outcome, will undergo an exploratory study to evaluate the effectiveness of algorithm based programming (Phase 1). Subsequently, patients undergoing STN DBS will be randomly allocated to algorithm based programming/ standard of care programming and after adequate stabilisation evaluated for motor improvement. They will be switched over to the alternative technique of programming and evaluated again after a similar period. Data regarding the time consumed, effectivity and several secondary endpoints will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of bilateral idiopathic Parkinson's disease
* Exhibit a UPDRS subset III score of ≥ 25 while in the preoperative medication off state
* Demonstrate an improvement of Parkinson's disease symptoms by ≥30% in the medication off state following a pre-operative levodopa challenge, as assessed by the UPDRS subset III score
* Possess the ability to comprehend the study's demands, treatment protocols, and procedures, and provide written informed consent before undergoing any study-specific tests or procedures

Exclusion Criteria:

* Patients with notable psychiatric conditions, including unrelated clinically substantial depression as assessed by the investigator, will be excluded from participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of efficacy between StimSearchTM-based programming and the best Standard of Care (SOC) based programming. | 4 weeks
  Unified Parkinson's disease rating scale scores (part III) will be used to evaluate this. Range (0-132) The lower the score indicates lesser severity of the disease and improved outcome.
Comparison of time required between StimSearch and SOC programming | 4 weeks
  Total time in minutes will recorded

SECONDARY OUTCOMES:
Comparison of volume of tissue activated (VTA) between StimSearch and SOC | 4 weeks
  The volume of tissue activated in cubic millimeter will be calculated.
Comparison of target volume between StimSearch and SOC | 4 weeks
  The target volume in cubic millimeter will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Doshi, MCh, Principal Investigator — Jaslok Hospital and Research Center
Locations (1):
- Jaslok Hospital And Research Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Malekmohammadi M, Mustakos R, Sheth S, Pouratian N, McIntyre CC, Bijanki KR, Tsolaki E, Chiu K, Robinson ME, Adkinson JA, Oswalt D, Carcieri S. Automated optimization of deep brain stimulation parameters for modulating neuroimaging-based targets. J Neural Eng. 2022 Jul 20;19(4):10.1088/1741-2552/ac7e6c. doi: 10.1088/1741-2552/ac7e6c. PMID 35790135
- [Result] Sasaki F, Oyama G, Sekimoto S, Nuermaimaiti M, Iwamuro H, Shimo Y, Umemura A, Hattori N. Closed-loop programming using external responses for deep brain stimulation in Parkinson's disease. Parkinsonism Relat Disord. 2021 Mar;84:47-51. doi: 10.1016/j.parkreldis.2021.01.023. Epub 2021 Jan 30. PMID 33556765
- [Result] Wenzel GR, Roediger J, Brucke C, Marcelino ALA, Gulke E, Potter-Nerger M, Scholtes H, Wynants K, Juarez Paz LM, Kuhn AA. CLOVER-DBS: Algorithm-Guided Deep Brain Stimulation-Programming Based on External Sensor Feedback Evaluated in a Prospective, Randomized, Crossover, Double-Blind, Two-Center Study. J Parkinsons Dis. 2021;11(4):1887-1899. doi: 10.3233/JPD-202480. PMID 34151855